CLINICAL TRIAL: NCT04140877
Title: Choroidal Changes Post Short Term Exposure To Virtual Reality Devices
Acronym: MIRABILE
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Strategy change
Sponsor: Visu, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: P/689/19/VU
Record Dates: First submitted 2019-10-21; First posted 2019-10-28 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-06

CONDITIONS: Myopia
Keywords: Choroidal thickness; Virtual reality
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Intervention Model Description: Randomized, contralateral eye study
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Visu OD, Control OS (Other): Contralateral eye study
  Interventions: Device: Visu
- Control OD, Visu OS (Other): Contralateral eye study
  Interventions: Device: Visu

INTERVENTIONS:
Device: Visu — An experimental (test) virtual reality display

SUMMARY:
This is a prospective, randomized, controlled, contralateral eye, clinical study. The objective of the study is to determine the impact of Virtual Reality (VR) usage on choroidal thickness when viewed through a test display compared to a control (standard) VR display. The hypothesis is that there will be less choroidal thinning in the eye viewing the test VR screen compared to the eye viewing the control VR screen.

ELIGIBILITY:
Key Inclusion Criteria:

* Is at least 13 years of age and has full legal capacity to volunteer;
* Has read and signed an information consent letter;
* Visual Acuity of +0.20 logMAR or better in each eye;
* Is willing and able to follow instructions and maintain the appointment schedule.

Key Exclusion Criteria:

* Is participating in any concurrent clinical or research study;
* Has any known active ocular disease and/or infection;
* Has a systemic condition that in the opinion of the investigator may affect a study outcome variable;
* Is amblyopic in either eye;
* Has a colour vision abnormality;
* Commonly experiences motion sickness.

Min Age: 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-07 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2021-01 (Estimated)

PRIMARY OUTCOMES:
Choroidal thickness | 2 hours

SECONDARY OUTCOMES:
Choroidal thickness | 3 months
Axial length | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Lyndon Jones, PhD, FCOptom, Principal Investigator — Centre for Ocular Research and Education

IPD SHARING:
Plan to Share IPD: No